CLINICAL TRIAL: NCT01892969
Title: Coagulation and Fibrinolysis in a Pediatric Insulin Titration Trial
Brief Title: Coagulation and Fibrinolysis in Pediatric Insulin Titration Trial (CAF-PINT)
Acronym: CAF-PINT
Status: Completed | Type: Observational
Sponsor: University of California, San Francisco (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Other Study IDs: A120253; 1R01HL114484-01A1 (NIH)
Record Dates: First submitted 2013-06-26; First posted 2013-07-08 (Estimated); Last update posted 2020-07-31 (Actual); Status verified 2020-07

CONDITIONS: Heart Failure; Respiratory Failure
MeSH Terms: conditions — Heart Failure; Respiratory Insufficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood Samples
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- HEART AND LUNG FAILURE: Patients with Heart failure or Respiratory Failure with Hyperglycemia

SUMMARY:
Project Summary We propose an ancillary study to The Heart and Lung Failure Pediatric Insulin Titration trial (HALF PINT), which is investigating the impact of normalizing blood glucose using insulin infusions on clinical outcomes among children with hyperglycemia and heart and lung failure. In this ancillary study, we will measure plasma levels of inflammatory, coagulation, and fibrinolysis proteins and genotype DNA for polymorphisms among patients enrolled in the HALF PINT trial. The results from this ancillary study will help us to understand potential mechanisms through which normalizing blood glucose provides benefit, which may lead to development of new therapeutic strategies in critically ill children

DETAILED DESCRIPTION:
ABSTRACT Hyperglycemia occurs frequently among critically ill children and is associated with increased morbidity and mortality. Approximately 25% of critically ill children with heart and lung failure (i.e., those receiving mechanical ventilation and/or inotropes) develop hyperglycemia within 24 hours of admission, and if the hyperglycemia is sustained (lasting for > 50% of PICU stay), it results in a 6-fold increase in the odds of mortality. Previous studies have demonstrated that tight glycemic control with insulin, aimed at achieving normoglycemia (TGC-NL) can result in improvement in mortality and morbidity in selected groups of critically ill patients with hyperglycemia. However, the precise mechanism by which TGC-NL leads to improvement in morbidity and mortality is not known. Hyperglycemia is known to result in a pro-thrombotic state via activation of coagulation and impairment of fibrinolysis. This pro-thrombotic, anti-fibrinolytic state, may lead to intravascular fibrin deposition and micro thrombi, which can be a key contributor to the pathogenesis of multi-organ failure. We propose to take advantage of The Heart and Lung Failure Pediatric Insulin Titration trial (HALF PINT) - an NHLBI-funded randomized, controlled trial designed to study the impact of TGC-NL on clinical outcomes among children with heart and lung failure - to investigate the effect of TGC-NL on inflammation, fibrinolysis, and coagulation and to determine the extent to which improvement in deranged coagulation and fibrinolysis by TGC-NL contributes to improvement in clinical outcomes. We propose to enroll 800 critically ill patients with hyperglycemia and heart and lung failure from the HALF PINT study. Since the parent trial will not collect any blood samples other than for confirmation of blood glucose, we will approach parents or surrogates of children enrolled in the HALF PINT trial and obtain informed consent for participation in this ancillary study. We will collect blood samples (3cc from children 2 years and younger, and 5ml from children 3 years and older) at Days 1, 3, and 5 after randomization. We will measure plasma levels of selected markers of coagulation and fibrinolysis and genotype DNA for polymorphisms in the corresponding genes. We will correlate changes over time in the biomarkers with allocation to treatment arm to test whether the beneficial effects of TGC-NL are achieved via normalization of coagulation and fibrinolysis. We will also genotype for tag SNPs in the corresponding genes and test for association of the plasma and genetic markers with clinical outcomes. The results from this study will provide mechanistic insights into the effect of TGC-NL on clinical outcome and could lead to the use of anti-inflammatory, anti-coagulant or pro-fibrinolytic agents as adjunctive therapies among select groups of critically ill children with hyperglycemia who may not be amenable to tight glucose control or are at higher risk of adverse clinical outcomes from a pro thrombotic environment. Results from this study may lead to identification of protein or genetic markers that will identify critically ill children most likely to benefit from existing anticoagulant therapies such as activated protein C.

ELIGIBILITY:
Inclusion Criteria:

All Patients enrolled in the HALF PINT trial

Exclusion Criteria:

Bleeding Diathesis as manifest by a Most Recent recorded International Normalized ratio (INR) >3

Ages: 14 Days to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients Enrolled in the Half Pint Trial to study the efficacy of Tight Glycemic control using Insulin on reducing organ failure and mortality among children with Heart and Lung Failure with Hyperglycemia
Sampling Method: Non-Probability Sample
Enrollment: 304 (Actual)
Dates: Start 2012-10; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Biomarkers of Thrombosis and Inflammation (Interleukin 6 (IL6) and Interleukin 8 (IL8) , Plasminogen Activator Inhibitor -1 (PAI-1)) | 4 days
  The researchers will measure IL-6, IL-8 and PAI-1 on patient plasma using a Luminex based multiplex array. All measurements are in pg/mL. The Slope of change in biomarkers from the time of start of insulin infusion to 2 and 4 days after start of insulin infusion will be used as the outcome measure.

SECONDARY OUTCOMES:
Number of participants with Development of Acute Lung Injury (ALI) | 28 days
  Acute Lung Injury (ALI) measured as hypoxemia with bilateral infiltrates

CONTACTS AND LOCATIONS:
Overall Officials: Anil Sapru, MD,MAS, Principal Investigator — University of California, Los Angeles
Locations (25):
- United States (25):
  - Children's Hospital of Los Angeles, Los Angeles, California
  - Mattel Children's Hospital (UCLA), Los Angeles, California
  - Children's Hospital and Research Center of Oakland, Oakland, California
  - Children's Hospital of Orange County, Orange, California
  - Children's Hospital Colorado - Denver, Aurora, Colorado
  - Yale - New Haven Children's Hospital, New Haven, Connecticut
  - Nemours/Alfred I. DuPont Hospital for Children, Wilmington, Delaware
  - Children's Healthcare of Atlanta (Emory), Atlanta, Georgia
  - Ann & Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois
  - University of Chicago Medicine Comer Children's Hospital, Chicago, Illinois
  - Indiana University Riley Hospital for Children, Indianapolis, Indiana
  - University of Louisville Children's Hospital, Louisville, Kentucky
  - Children's Hospital of Boston, Boston, Massachusetts
  - C.S. Mott Children's Hospital - Michigan, Ann Arbor, Michigan
  - St. Louis Children's Hospital, St Louis, Missouri
  - Dartmouth Hitchcock Medical Center, Manchester, New Hampshire
  - Women and Children's Hospital of Buffalo, Buffalo, New York
  - Cohen Children's Medical Center of NY/ North Shore LIJ, New Hyde Park, New York
  - Maria Fareri Children's Hospital at Westchester Medical Center, Valhalla, New York
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - PennState Hershey Medical Center, Hershey, Pennsylvania
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Medical City Children's Dallas, Dallas, Texas
  - Children's Medical Center Dallas, Dallas, Texas
  - Primary Children's Medical Center, Salt Lake City, Utah

REFERENCES:
- [Derived] Zinter MS, Markovic D, Asaro LA, Nadkarni VM, McQuillen PS, Sinha P, Matthay MA, Jeschke MG, Agus MSD, Sapru A; CAF-PINT Investigators of the PALISI Network. Tight Glycemic Control, Inflammation, and the ICU: Evidence for Heterogeneous Treatment Effects in Two Randomized Controlled Trials. Am J Respir Crit Care Med. 2023 Apr 1;207(7):945-949. doi: 10.1164/rccm.202210-1988LE. No abstract available. PMID 36656551